CLINICAL TRIAL: NCT05963048
Title: Comparative Study About Effect of Rituximab Versus IL-6 Inhibitor in Induction of Remission in Active ILD in Scleroderma Patients
Brief Title: Rituxmab Versus IL-6 in Treating ILD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Scleroderma
Record Dates: First submitted 2022-12-25; First posted 2023-07-27 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Interstitial Lung Disease; Scleroderma
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Diffuse | interventions — Rituximab; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: participant and outcome assrssor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituxmab (Experimental): 1000 mg Rituxmab IV infusion at 1st day then after 15 weeks then after 6 months for 1 year
  Interventions: Drug: Rituximab
- IL-6 inhibitor (Experimental): 6 mg/kg IV infusion every month not exceed 600 mg for 1 year
  Interventions: Drug: IL6 inhibitor

INTERVENTIONS:
Drug: Rituximab — IV infusion 1000 mg
  Other Names: Rituxan
  Arms: Rituxmab
Drug: IL6 inhibitor — 6 mg/kg I V infusion monthly
  Other Names: Actemra
  Arms: IL-6 inhibitor

SUMMARY:
All SSc patients should know if they have been diagnosed with interstitial lung disease, or pulmonary hypertension and keep results from his/her last pulmonary function test, chest imaging, echocardiogram and stress test

DETAILED DESCRIPTION:
All SSc patients should know if they have been diagnosed with interstitial lung disease, or pulmonary hypertension and keep results from his/her last pulmonary function test, chest imaging, echocardiogram and stress test Diffuse infiltrative lung disease (ILD): progressive shortness of breath is the most frequently presentation going to ER pulmonary unit first. It should be considered in case of persistent dry cough or dyspnea, which should be looked for in any patient with SSc. an etiological assessment must be conducted in order not to mistakenly attribute ILD to the SSc.

ELIGIBILITY:
Inclusion Criteria:

* active ILD scleroderma

Exclusion Criteria:

* abnormal liver enzymes renal impairment neutropenia <1000 cells/mm3 thrombocytopenia < 50,000 cells/mm3

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
forced vital capacity | 6 months
  pulmonary function test

SECONDARY OUTCOMES:
computed tomography chest | 1 year
  imaging
modified rodnan skin score | 6 months
  skin score

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hassanien, MD, Principal Investigator — Assiut University
Locations (1):
- Manal Hassanien, Asyut, Yes, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after finishing
Supporting Information: Study Protocol, CSR
Time Frame: one year
Access Criteria: after finishing the study